CLINICAL TRIAL: NCT03222817
Title: HPV Self-Sampling for Cervical Cancer Screening Among Transgender Men and Transmasculine Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Julia Seay, Research Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20170329
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Self-sampling (Experimental): All participants will receive HPV self-sampling. HPV self-sampling allows an individual to screen themselves for cervical cancer in private, using a device that is similar to a tampon.
  Interventions: Behavioral: HPV self-sampling

INTERVENTIONS:
Behavioral: HPV self-sampling — Participants will be provided with education regarding cervical cancer screening, as well as instructions regarding how to use the HPV self-sampler. Participants will also receive referrals to trans-competent healthcare providers for follow-up screening and care.

SUMMARY:
The proposed study will examine the implementation of a Human Papillomavirus (HPV) self-sampling intervention for unscreened and under-screened transgender men and transmasculine individuals living in South Florida. The study will enroll participants to receive this cervical cancer screening intervention in community venues. The purpose of this study is to pilot the self-sampler for feasibility and acceptability within this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as transgender male or as transmasculine

  * Assigned female sex at birth
  * English speaking
  * ages 25-65 years
  * report not having had a pap smear in the last three years
  * if age 30 and over, report not having a Pap smear/HPV co-test in the past 5 years

Exclusion Criteria:

* • Those who report having had a hysterectomy

  * Those who report having history of cervical cancer
  * Adults unable to consent
  * Those who are pregnant
  * Prisoners

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be assigned female sex at birth and identify as transgender male or transmasculine.
Enrollment: 10 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Acceptability of HPV self-sampling Questionnaire | This questionnaire will be administered immediately after participants self-sample
  This questionnaire, designed with substantial input from community partners, will gauge how acceptable the participants find HPV self-sampling through both closed and open-ended questions regarding ease of use, preference of self-sampler vs. physician-collected Pap smear, as well as open-ended inquiries regarding the self-sampling process.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No